CLINICAL TRIAL: NCT04560270
Title: KRAS (Kirsten Rat Sarcoma) Mutant CIrculating Tumor DNA for Monitoring Response to First Line Chemotherapy in Locally Advanced and Metastatic PANcreatic Cancer
Brief Title: CIrculating Tumor DNA for Monitoring Response to First Line Chemotherapy in Unresectable PANcreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KRASCIPANC
Record Dates: First submitted 2020-09-05; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer; Circulating Tumor DNA; KRAS Mutation-Related Tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only arm (Experimental): Blood samples to analyze ctDNA
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Blood samples to determine ctDNA levels during chemotherapy

SUMMARY:
With an incidence of more than 11,600 new cases per year in France and an annual number of deaths close to the incidence rate, adenocarcinoma of the pancreas is a public health problem.

The aim of this study is to assess the predictive value of response to the 1st line of chemotherapy of mutated KRAS ctDNA (circulating tumor DNA) in unresectable metastatic or locally advanced pancreatic adenocarcinomas.

DETAILED DESCRIPTION:
With an incidence of more than 11,600 new cases per year in France and an annual number of deaths close to the incidence rate, adenocarcinoma of the pancreas is a public health problem especially since there is a significant increase in its incidence. incidence (+ 417% between 1980 and 2012).

Most often diagnosed late, pancreatic adenocarcinoma is managed at a metastatic stage in 60 to 70% of cases with a very poor prognosis (8.7 to 11.1 months median survival with current chemotherapies). The first line of chemotherapy therefore represents a major issue in the management of these unresectable patients. There are few predictive markers of response to chemotherapy in pancreatic adenocarcinoma. It is conventionally evaluated by scanner every 2 to 3 months. The response to chemotherapy is associated with a good prognosis while non-response has a poor prognosis and requires a 2nd line of treatment if the patient is able to receive it.

A KRAS mutation is present in approximately 70-90% of pancreatic adenocarcinomas. Its research on tissue sampling (fine needle aspiration or anatomo-pathological specimen) is not carried out routinely because no prognostic or predictive value of KRAS mutations has been demonstrated. New high-throughput DNA sequencing techniques have been developed and now allow a blood sample to detect and quantify circulating tumor DNA (ctDNA), including KRAS mutations.

Very few studies have investigated the change in cDNA levels during 1st line chemotherapy in unresectable pancreatic adenocarcinoma.

The aim of this study is to assess the predictive value of response to the 1st line of chemotherapy of mutated KRAS cDNA in unresectable metastatic or locally advanced pancreatic adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Proven pancreatic adenocarcinoma (histology or cytology)
* Metastatic or locally advanced unresectable
* With thoraco-abdomino-pelvic scanner less than a month old
* Chemotherapy treatment regardless of the protocol
* Patients benefiting from a Social Security scheme or benefiting through the intermediary of a third party
* Informed consent signed by the patient after clear and fair information about the study

Exclusion Criteria:

* Linguistic or psychological refusal or inability to understand and / or sign the informed consent
* History of cancer in the 5 years preceding inclusion
* Patient who has already received chemotherapy or radiotherapy for pancreatic cancer.
* Immediately resectable tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Correlation of the ctDNA level to the response to chemotherapy | 3 months
  Response to chemotherapy was evaluated with RECIST criteria 1.1 on the first CT scan

SECONDARY OUTCOMES:
Overall survival | 6 months after last patients inclusion
  Correlation between variation of ctDNA and overall survival
Progression free survival | 6 months after last patients inclusion
  Correlation between variation of ctDNA and progression free survival

REFERENCES:
- [Derived] Evrard C, Ingrand P, Rochelle T, Martel M, Tachon G, Flores N, Randrian V, Ferru A, Haineaux PA, Goujon JM, Karayan-Tapon L, Tougeron D. Circulating tumor DNA in unresectable pancreatic cancer is a strong predictor of first-line treatment efficacy: The KRASCIPANC prospective study. Dig Liver Dis. 2023 Nov;55(11):1562-1572. doi: 10.1016/j.dld.2023.03.011. Epub 2023 Jun 10. PMID 37308396